CLINICAL TRIAL: NCT05513859
Title: Towards In-Vivo, Intraoperative Image Guided Brain Tumor Margin Assessment With Quantitative Oblique Back Illumination Microscopy
Brief Title: Investigational Imaging Technique During Brain Surgery
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Temporarily Closed
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Jeffrey James Olson, Principal Investigator, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY00004168; NCI-2022-06212 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00004168 (Other: Emory University Hospital/Winship Cancer Institute); WINSHIP5571-22 (Other: Emory University Hospital/Winship Cancer Institute); P30CA138292 (NIH)
Record Dates: First submitted 2022-08-22; First posted 2022-08-24 (Actual); Last update posted 2025-06-03 (Actual); Status verified 2025-05

CONDITIONS: Astrocytoma; Glioblastoma; Oligodendroglioma
MeSH Terms: conditions — Astrocytoma; Glioblastoma; Oligodendroglioma | interventions — Craniotomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Diagnostic (qOBM) (Experimental): Patients undergo craniotomy with intraoperative ex vivo and in situ tumor assessment with qOBM. Patients then undergo postoperative exam with CT or MRI any of days 1-5 after surgery.
  Interventions: Procedure: Craniotomy; Device: Quantitative Oblique Back-Illumination Microscopy

INTERVENTIONS:
Procedure: Craniotomy — Undergo craniotomy
  Other Names: Open Craniotomy
Device: Quantitative Oblique Back-Illumination Microscopy — Undergo intraoperative microscopy utilizing qOBM
  Other Names: qOBM

SUMMARY:
This early phase I trial tests the safety and reliability of an investigational imaging technique called quantitative oblique back illumination microscopy (qOBM) during brain surgery for detecting brain tumors and brain tumor margins in patients with glioblastoma, astrocytoma, or oligodendroglioma. Surgical margins refer to the edge or border of the tissue removed in cancer surgery. qOBM may be able to assess and reveal brain tumor surgical margins in a more safe and reliable manner.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To perform a first-in-human study to assess the ability of a quantitative oblique back illumination microscopy (qOBM) handheld device to safely and reliably image brain tumor pathology intraoperatively in-situ and in-vivo.

SECONDARY OBJECTIVES:

I. To characterize the biophysical and structural features that enable detection of bulk tumor and tumor margins, including infiltrative disease, with qOBM.

II. To develop qOBM imaging probes with multimodal capabilities (analog black and white and color imaging, fluorescent imaging) and with the potential to clearly reveal brain tumor margins ex vivo and in vivo during neurosurgical procedures.

OUTLINE:

Patients undergo craniotomy with intraoperative ex vivo and in situ tumor assessment with qOBM. Patients then undergo postoperative exam with computed tomography (CT) or magnetic resonance imaging (MRI) any of days 1-5 after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 18 years
* Craniotomy is indicated for tumor management
* Surgery planned for 14 or fewer days from enrollment
* Evidence of a personally signed informed consent indicating that the subject is aware of the neoplastic nature of the disease and has been informed of the procedures to be followed, the experimental nature of the device evaluation, alternatives, potential risks and discomforts, potential benefits, and other pertinent aspects of study participation.
* A newly discovered brain lesion requiring surgery who imaging is consistent with a new glioblastoma, astrocytoma, or oligodendroglioma or with a progressive histologically proven glioblastoma, astrocytoma, or oligodendroglioma whose management required surgery.

Exclusion Criteria:

An individual who meets any of the following criteria will be excluded from participation in this study:

* Patients who are undergoing needle biopsy only
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2024-03-11 (Actual); Primary Completion 2026-06-28 (Estimated); Study Completion 2027-06-23 (Estimated)

PRIMARY OUTCOMES:
Incidence of Adverse Events | Up to 3 years
  Adverse events will be assessed and graded according to the Common Terminology Criteria for Adverse Events version 5.0. Summary statistics will be reported for categorical variables using descriptive statistics. Patient demographics will be summarized descriptively. 95% confidence intervals will be reported, unless otherwise specified. All tests will be two-sided.
Reliability of Quantitative Oblique Back Illumination Microscopy Device Determined by Frequency Distribution | Up to 3 years
  Robustness will be defined as the device's ability to clearly reveal relevant cellular and subcellular histological structures that can lead to clinically actionable outcomes, is determined. Using standard clinical techniques such as loupe magnification, surgical microscopy, histology, intraoperative ultrasound, and postoperative magnetic resonance imaging (MRI) as general points of historical reference.
  Summary statistics will be reported for categorical variables using descriptive statistics measures of frequency. Patient demographics will be summarized descriptively. All tests will be two-sided.
Reliability of Quantitative Oblique Back Illumination Microscopy Device Determined by Standard Deviation | Up to 3 years
  Robustness will be defined as the device's ability to clearly reveal relevant cellular and subcellular histological structures that can lead to clinically actionable outcomes, is determined. Using standard clinical techniques such as loupe magnification, surgical microscopy, histology, intraoperative ultrasound, and postoperative magnetic resonance imaging (MRI) as general points of historical reference.
  Summary statistics will be reported for categorical variables using standard deviation.Patient demographics will be summarized descriptively. 95% confidence intervals will be reported, unless otherwise specified. All tests will be two-sided.
Reliability of Quantitative Oblique Back Illumination Microscopy Device Determined by Central Tendency | Up to 3 years
  Robustness will be defined as the device's ability to clearly reveal relevant cellular and subcellular histological structures that can lead to clinically actionable outcomes, is determined. Using standard clinical techniques such as loupe magnification, surgical microscopy, histology, intraoperative ultrasound, and postoperative magnetic resonance imaging (MRI) as general points of historical reference.
  Summary statistics will be reported for categorical variables using descriptive statistics measures of central tendency. Patient demographics will be summarized descriptively. 95% confidence intervals will be reported, unless otherwise specified. All tests will be two-sided.
Reliability of Quantitative Oblique Back Illumination Microscopy Device Determined by Measures of Position | Up to 3 years
  Robustness will be defined as the device's ability to clearly reveal relevant cellular and subcellular histological structures that can lead to clinically actionable outcomes, is determined. Using standard clinical techniques such as loupe magnification, surgical microscopy, histology, intraoperative ultrasound, and postoperative magnetic resonance imaging (MRI) as general points of historical reference.
  Summary statistics will be reported for categorical variables using descriptive statistics interquartile range. Patient demographics will be summarized descriptively. 95% confidence intervals will be reported, unless otherwise specified. All tests will be two-sided.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey J. Olson, MD, Principal Investigator — Emory University Hospital/Winship Cancer Institute
Locations (1):
- Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia, United States